CLINICAL TRIAL: NCT00003515
Title: Phase II Study of Antineoplastons A10 and AS2-1 in Patients With Primitive Neuroectodermal Tumor Outside the Central Nervous System
Brief Title: Antineoplaston Therapy in Treating Patients With Metastatic, Recurrent, or Refractory Primitive Neuroectodermal Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066558; BC-PN-02 (Other: Burzynski Research Institute)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Primitive Neuroectodermal Tumor
Keywords: Metastatic Primitive Neuroectodermal Tumor; Recurrent Primitive Neuroectodermal Tumor; Refractory Primitive Neuroectodermal Tumor
MeSH Terms: conditions — Neuroectodermal Tumors, Primitive | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Patients With Metastatic, Recurrent, or Refractory Primitive Neuroectodermal Tumors will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
Current therapies for Metastatic, Recurrent, or Refractory Primitive Neuroectodermal Tumors provide very limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of Metastatic, Recurrent, or Refractory Primitive Neuroectodermal Tumors.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on patients with Metastatic, Recurrent, or Refractory Primitive Neuroectodermal Tumors.

DETAILED DESCRIPTION:
OVERVIEW: This is a single arm, open-label study in which patients with Metastatic, Recurrent, or Refractory Primitive Neuroectodermal Tumors receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues up to12 months in the absence of disease progression or unacceptable toxicity.

OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in patients with Metastatic, Recurrent, or Refractory Primitive Neuroectodermal Tumors, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in patients with Metastatic, Recurrent, or Refractory Primitive Neuroectodermal Tumors.
* To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed incurable primitive neuroectodermal tumors outside the central nervous system that are unlikely to respond to existing therapy, meeting 1 of the following criteria:

  * Metastatic disease
  * Progressive, recurrent, or refractory disease after initial therapy, including surgery, chemotherapy, and/or radiotherapy
* Measurable disease by MRI or CT scan
* Tumor must be at least 2 cm

PATIENT CHARACTERISTICS:

Age:

* 6 months and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC at least 2,000/mm^3
* Platelet count at least 50,000/mm^3

Hepatic:

* No hepatic insufficiency
* Bilirubin no greater than 2.5 mg/dL
* SGOT and SGPT no greater than 5 times upper limit of normal

Renal:

* No renal insufficiency
* Creatinine no greater than 2.5 mg/dL
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No uncontrolled hypertension
* No history of congestive heart failure
* No history of other cardiovascular conditions that contraindicate high dosages of sodium

Pulmonary:

* No serious lung disease, such as chronic obstructive pulmonary disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No active infection
* No nonmalignant systemic disease
* Not a high medical or psychiatric risk

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy
* No concurrent immunomodulating agents

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)

Endocrine therapy:

* Concurrent corticosteroids allowed

Radiotherapy:

* See Disease Characteristics
* At least 8 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics
* Recovered from prior surgery

Other:

* Prior cytodifferentiating agents allowed
* No prior antineoplastons
* No other concurrent antineoplastic agents

Ages: 6 Months to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 1996-12-12 (Actual); Primary Completion 1997-01-03 (Actual); Study Completion 1997-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com